

# Non-Interventional Study (NIS) Protocol

| Document Number: | c38660249-01 |
|---|---|
| BI Study Number: | 1237-0110 |
| BI Investigational Product(s): | Spiolto Respimat |
| Title: | Effectiveness of Maintenance Treatment with Tiotropium + Olodaterol in Comparison to Inhaled Corticosteroids + Long-acting β2 agonists in COPD patients in Taiwan: a non-interventional study based on the Taiwan National Health Insurance (NHI) data. |
| Brief lay title: | Effectiveness of Tiotropium + Olodaterol versus ICS+LABA among COPD patients in Taiwan |
| Protocol version identifier: | 1.0 |
| Date of last version of protocol: | Not applicable |
| PASS: | No |
| EU PAS register<br>number: | Study not registered |
| Active substance: | Tiotropium + Olodaterol (R03AL06) |
| Medicinal product: | Spiolto Respimat |
| Product reference: | BC26735443 |
| Procedure number: | Not applicable |
| Marketing authorisation holder(s): | Boehringer Ingelheim International GmbH |
| Joint PASS: | No |
| Research question and objectives: | To compare the risk of exacerbations between initiators of Tiotropium / Olodaterol (Tio/Olo) and inhaled corticolsteroids / long-acting $\beta$ 2-agonists (ICS/LABA) in a real world setting |
| Author: | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Marketing authorisation holder(s): | Boehringer Ingelheim International GmbH |
|---|---|
| MAH contact person: | Not applicable |
| EU-QPPV: | EU-QPPV: Not applicable |
| Signature of EU-QPPV: | Not applicable |
| <b>Date:</b> 23 May 2022 | |
| Proprietary confidential information © 2022 Boehringer Ingelheim Group of companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission | |

NIS Protocol BI Study Number: 1237-0110  c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

## 1. TABLE OF CONTENTS

| TITLI | E PAGI | E1 |
|-------|---------|----------------------------------|
| 1. | TABLE | E OF CONTENTS |
| 2. | LIST C | F ABBREVIATIONS5 |
| 3. | RESPC | NSIBLE PARTIES5 |
| 4. | ABSTF | PACT |
| 5. | AMEN | DMENTS AND UPDATES19 |
| 6. | MILES | TONES |
| 7. | RATIO | NALE AND BACKGROUND21 |
| 8. | RESEA | ARCH QUESTION AND OBJECTIVES22 |
| | | ARCH METHODS23 |
| 9.1 | STU | DY DESIGN23 |
| 9.2 | SET | TING |
| 9.2 | 2.1 | Study sites |
| 9.2 | 2.2 | Study population |
| 9.2 | 2.3 | Study visits |
| 9.2 | 2.4 | Study discontinuation |
| 9.3 | VAI | RIABLES24 |
| 9.3 | 3.1 | Exposures |
| 9.3 | 3.2 | Outcomes |
| | 9.3.2.1 | Primary outcomes |
| _ | 9.3.2.2 | Secondary outcomes |
| 9.3 | 3.3 | Covariates |
| 9.4 | | TA SOURCES28 |
| 9.5 | | TDY SIZE29 |
| 9.6 | | TA MANAGEMENT29 |
| 9.7 | | TA ANALYSIS29 |
| 9.′ | 7.1 | Main analysis29 |
| | 7.3 | Safety Analysis 31 |
| 9.8 | _ | ALITY CONTROL 31 |
| 9.9 | | ITATIONS OF THE RESEARCH METHODS |
| 9.10 | | HER ASPECTS |
| 9. | 10.1 | Data quality assurance |

| NIS | S Proto | ocol | |
|------|---------|---------|-----------|
| BI S | Study | Number: | 1237-0110 |

 c38660249-01

| Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated | |
|---|---|
| 9.10.2 Study records | 32 |
| 9.10.2.1 Source documents | 32 |
| 9.10.2.2 Direct access to source data and documents | 33 |
| 10. PROTECTION OF HUMAN SUBJECTS | 34 |
| 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT | 2.4 |
| 10.2 STATEMENT OF CONFIDENTIALITY | |
| 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 35 |
| 11.1 DEFINITIONS OF ADVERSE EVENTS | 35 |
| 11.2 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AN REPORTING | |
| 11.3 REPORTING TO HEALTH AUTHORITIES | 35 |
| 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 36 |
| 13. REFERENCES | 37 |
| 13.1 PUBLISHED REFERENCES | 37 |
| 13.2 UNPUBLISHED REFERENCES | 37 |
| ANNEX 1. LIST OF STAND-ALONE DOCUMENTS | 38 |
| ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 39 |
| ANNEX 3. ADDITIONAL INFORMATION | 46 |
| ANNEX 4 REVIEWERS AND APPROVAL SIGNATURES | 47 |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

## 2. LIST OF ABBREVIATIONS

AE Adverse Event

CA Competent Authority
CI Confidence Interval

COPD Chronic Obstructive Pulmonary Disease

ENCePP European Network of Centres for

Pharmacoepidemiology and Pharmacovigilance

GPP Good Pharmacoepidemiology Practice GVP Good Pharmacovigilance Practices

ICS Inhaled corticolsteroids

IEC Independent Ethics Committee
 IRB Institutional Review Board
 LABA Long-acting β2-agonists

LAMA Long-acting muscarinic antagonists
MAH Marketing Authorization Holder
NHI Taiwan National Health Insurance

NIS Non-Interventional Study

Olo Olodaterol

PASS Post-Authorization Safety Study

SAE Serious Adverse Event

Tio Tiotropium

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

# 3. RESPONSIBLE PARTIES

| BI NIS Lead (Scientific) BI NIS Lead (Operation) |
|---------------------------------------------------|
| BI NIS Lead (Operation) |
| BI NIS Lead (Operation) |
| BI NIS Lead (Operation) |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

## 4. ABSTRACT

COPD is a leading cause of morbidity and mortality throughout the world. Long-acting bronchodilator medications, which include long-acting β2-agonists (LABAs) and the long-acting muscarinic antagonists (LAMAs) such as tiotropium, are the central maintenance therapy to the management of COPD, with inhaled corticosteroids (ICSs) added with increasing severity. The up-to-date GOLD guideline recommends to initiate ICS/LABA in patients with high blood eosinophils level and frequent exacerbation history[P21-01394]. However, ICS containing therapy has been widely used inappropriately in real world practice.

The role of ICS in COPD has been debated for decades and studies have been conducted to investigate the effect of ICS-containing therapy in patients with COPD. INSPIRE [P07-11820] study indicated that ICS/LABA and tiotropium showed similar effects on the reduction of exacerbations, while the risk of pneumonia was higher in the ICS/LABA group. And the FLAME [P16-05628] study showed LAMA/LABA was superior to ICS/LABA in terms of exacerbation prevention, while in some newly published data focusing on FDC triple therapy showing reversed results.

With more and more fixed dose combination medications, i.e. LAMA/LABA, ICS/LABA/LAMA, approved and prescribed in recent years, it is of clinical interests to understand the effectiveness and safety profile of these therapies in real world settings.

The aim of this real world study is to assess effectiveness and safety profile between tiotropium/olodaterol (Tio/Olo) and ICS/LABA. The primary outcome of the study will be risk of moderate or severe COPD exacerbations. Other outcomes include time to ICS/LABA/LAMA escalation, rate of escalation to triple therapy, pneumonia and rescue medication use.

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelhein | n | | |
| Name of finished mo<br>product:<br>Spiolto Respimat | edicinal | | |
| Name of active ingre<br>Tiotropium + Olodate<br>{R03AL06} | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| Title of study: | Effectiveness of Maintenance Treatment with Tiotropium + Olodaterol in Comparison to Inhaled Corticosteroids + Long-acting β2 agonists in COPD patients in Taiwan: a non-interventional study based on the Taiwan National Health Insurance (NHI) data | | |
| Rationale and background: | world. Long-ac acting β2-agoni (LAMAs) such management of increasing seve initiate ICS/LA frequent exacer therapy has been conducted patients with CICS/LABA and exacerbations, group. And the superior to ICS some newly pureversed results. With more and LAMA/LABA, years, it is of cl profile of these. The aim of this results outcome of the serversed results. | ling cause of morbidity and morbiding bronchodilator medication ists (LABAs) and the long-acting as tiotropium, are the central in a COPD, with inhaled corticoste crity. The up-to-date GOLD guida. BA in patients with high blood rebation history [P21-01394]. Here is in COPD has been debated for a to investigate the effect of ICS OPD. INSPIRE [P07-11820] and tiotropium showed similar effect while the risk of pneumonia was FLAME [P16-05628] study and FLABA in terms of exacerbation blished data focusing on FDC to a superior of the control of th | s, which include longing muscarinic antagonists naintenance therapy to the eroids (ICSs) added with deline recommends to leosinophils level and lowever, ICS containing in real world practice. If decades and studies have decades and studies have decades and studies have decades and studies have decades and studies have decades on the reduction of less higher in the ICS/LABA howed LAMA/LABA was on prevention, while in riple therapy showing decades and safety profile decades and safety profile decades. |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | 1 | | |
| Name of finished medicinal | | | |
| product: | Michigan | | |
| Spiolto Respimat | | | |
| Name of active ingre<br>Tiotropium + Olodate | | | |
| {R03AL06} | 101 | | |
| (Rosando) | | | |
| Protocol date: | Study | Version/Revision: | Version/Revision date: |
| | number: | | |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| | escalation, rate medication use | of escalation to triple therapy, | pneumonia and rescue |
| Research question | Primary objecti | ive· | |
| and objectives: | • | | ware CODD evacerbations |
| | To compare time to the first moderate or severe COPD exacerbations between initiators of Tiotropium / Olodaterol (Tio/Olo) and inhaled | | |
| | corticolsteroids / long-acting β2-agonists (ICS/LABA) after entry | | |
| | between 1st January 2014 and 31st December 2019 | | |
| | Secondary objectives: | | |
| | <ul> <li>To compare time to escalation to triple therapy between initiators of<br/>Tio/Olo and ICS/LABA;</li> </ul> | | |
| | <ul> <li>To compare the rate of escalation to triple therapy between initiators<br/>of Tio/Olo and ICS/LABA;</li> </ul> | | |
| | _ | ompare the time to first hospitalization for community-acquired monia between initiators of Tio/Olo and ICS/LABA; | |
| | | pare the number of prescriptions of rescue medication between s of Tio/Olo and ICS/LABA | |
| | To compare exacerbation | compare the annualized rate of moderate or severe COPD | |
| | | l of between 1st January 2014 a | nd 31st December 2019 |
| | | ry objectives above | nd 31st December 2017 |
| Study design: | | e a non-interventional cohort st | tudy based on existing data |
| | (NISed). | | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | 1 | | |
| Name of finished me product: Spiolto Respimat | edicinal | | |
| Name of active ingredient: Tiotropium + Olodaterol {R03AL06} | | | |
| (ROSTEOO) | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| Population: | Inclusion criter | ia: | |
| | LABA/ICS<br>December 2 | | |
| | _ | O years on the index date one diagnosis of COPD at any time prior to or on the index one year of continuous medical and health insurance plan prior ex date will be required to allow for a look-back period for intest and identification of new use of the study drugs; | |
| | to the index<br>the covarian | | |
| | 5. At least one | e record in the health insurance | system database; |
| | Exclusion criter | ria: | |
| | | LAMA/LABA, ICS/LABA, or rm for one year prior to the inde | |
| | 2. Individuals | with asthma, allergic rhinitis, l | ung cancer, interstitial lung |
| | disease, or | lung transplant identified at any | time prior to the index date; |
| Variables: | Exposures: | • | |
| | Exposure of this study is defined as new initiation of Tiotropium/Olodaterol, or ICS/LABA during the study period. | | |
| | Outcomes: | | |
| | Primary outcon | | |
| | • Time to the entry | | |
| | _ | comes: le therapy escalation after entry ate of triple therapy initiation; | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| | | | _ |
|---|---|---|---|
| Name of company: | | | |
| Boehringer Ingelhein | ı | | |
| Name of finished me product: Spiolto Respimat | edicinal | | |
| Name of active ingredient: Tiotropium + Olodaterol {R03AL06} | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| | pneumonia Annualized as: annualized as: annualized (calculated COPD exace exacerbation Covariates: Demographic Sex Age Calendar y Season of i Additional, the measured duri Specific prev LAMA is LABA is ICS more | I rate of prescriptions of rescripted rate=number of prescriptions per patient of prescriptions per patient rate of moderate or severe (as: annualized rate=number cerbations/total patient year as ons per patient year) characteristics and cohort entry and and the characteristics and cohort entry and the characteristics and char | ue medications (calculated ions/total patient year at t year); COPD exacerbation of moderate or severe at risk=number of htty information: mmer, fall) |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished me product: Spiolto Respimat | dicinal | | |
| Name of active ingre<br>Tiotropium + Olodate<br>{R03AL06} | | | |
| Protocol date: | Study | Version/Revision: | Version/Revision date: |
| 23 May 2022 | number:<br>1237-0110 | 1.0 | NA |
| | Use of other re | espiratory drugs | |
| | Mucoly | tics | |
| | > Theophy | ylline | |
| ➤ Short-ac | | eting beta-agonists | |
| | ➤ Short-ac | cting muscarinic antagonists | |
| | both 12 m categorize All ex An or any fr an an Hosp prima diagn Number of | of hospitalizations caused by | ere) is code for COPD in ral corticosteroid or ions (Moderate) om visits with a |
| | > 0;<br>> 1;<br>> 2+; | 12 months prior to the index of all-cause hospitalizations in e: | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of company: | | | |
|---|---|---|---|
| Name of finished medicinal product: Spiolto Respimat | | | |
| Name of active ingre<br>Tiotropium + Olodate<br>{R03AL06} | | | |
| Protocol date: | Study | Version/Revision: | Version/Revision date: |
| | number: | | |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| | <ul> <li>Cerel</li> <li>Diabe</li> <li>Chro</li> <li>Pneu</li> <li>Canc</li> <li>Cirrh</li> <li>Charlson</li> <li>History of or on the dispensing</li> <li>Cardinantian intrate heart</li> <li>Lipid</li> <li>Blood</li> <li>Antic</li> <li>Antic</li> </ul> | iovascular disease provascular disease etes nic kidney disease monia er osis Comorbidity Index (CCI) f medications dispensed in index date will be identifie g history: iovascular drugs: ypertensives rrhythmics tes failure medications d-lowering medications d glucose-lowering medicat coagulants and antiplatelet a piotics meoplastic agents | d from the pharmacy |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelhein | 1 | | |
| Name of finished me product: Spiolto Respimat | edicinal | | |
| Name of active ingre<br>Tiotropium + Olodate<br>{R03AL06} | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| Data sources: | Data used in this study will come from the Taiwan National Health Insurance (NHI) claims data between 2014 and 2019. Data sources include Taiwan NHI, Taiwan cancer registry (TCR) and Taiwan Mortality Data. Taiwan Department of Statistics, Ministry of Health and Welfare is the unit designated by the government to manage health and social welfare statistical databases, and to develop data platform for academic research. Through the services provided by the Health and Welfare Data Science Center (HWDSC) of the Department of Statistics, researchers may access a wide range of health and welfare data, including claims, mortality (with cause of death) and Taiwan Cancer Registry (TCR). The HWDSC staff encrypt the national ID for all individuals according to a secure encryption algorithm that is not made known to the public. The encrypted ID is unique for all individuals and will be used for linkage between databases. | | |
| | Taiwan Nation publicly funderesidents. Heat coverage is martaiwan contrataiwan to prolocations of heat Taiwan. Salar premium calcusocioeconomic Related Group | ional Health Insurance (NHI) started in 1995 and is a added single payer health insurance program for all fealth insurance for individuals is required by law and more than 99%. The majority of healthcare providers in tract with the National Health Insurance Agency in provide a wide range of medical services. Geographic health care claims are broadly classified into 6 regions in lary range, which serves as the basis for enrollees' alculation, can serve as a proxy indicator for mic status. Bundled payment according to the Diagnosistup system only applies in limited number of disease therefore detailed drug use information during | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | 1 | | |
| Name of finished me product: Spiolto Respimat | | | |
| Name of active ingre<br>Tiotropium + Olodate<br>{R03AL06} | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| | source is the leading of the important for International Commodification (switched to Inclinical modificate column position (No document accessed by Position). | data | e, which is particularly WHI claims were based on th revision, clinical d of 2015, and then Disease, tenth revision, after 2016. Specific NHI in_TW_NHI_20210824" tial and only can be |
| | status, and dea<br>of Household<br>certificates are<br>Ministry of Ho<br>death and mai<br>was coded in the<br>10-CM formate<br>death files in year | the household registration system in Taiwan maintain birds tus, and death information and is administrated by the I Household Registration, Ministry of the Interior. Death tificates are collected through this system and transferrentistry of Housing and Works (MOHW) for coding of cath and maintenance of the mortality database. The causes coded in the ICD-9-CM format from 1990 to 2009, are CM format from 2010 to 2019. This study will use the ath files in years 2012-2019, primarily focusing on the outh of study subjects. | |
| | In Taiwan, the<br>1979. Since the<br>the "20 items<br>(including can<br>from hospitals<br>country. Reco<br>method of dia | e population-based cancer regien, the registry collected bas short-form system," on incid acer-in-situ) within one year as with more than 50-bed capa rded items include date of big gnosis, cancer site and morpl death. From 2002 onward, a | ic information, referred to<br>ent cancer cases<br>after the initial diagnosis<br>city throughout the<br>rth, gender, time and<br>hology, treatment |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of company: | - | Boehringer Ingelheim International GmbH of | |
|---|---|---|---|
| Boehringer Ingelhein | 1 | | |
| Name of finished medicinal product: Spiolto Respimat | | | |
| Name of active ingredient: Tiotropium + Olodaterol {R03AL06} | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| | established to collect more detailed information of cancer staging, treatment and follow-up data from hospitals with more than 500 new cancer cases diagnosed annually. The number of recorded items increased from 20 to 65 in 2002, further to 95 in 2007, and to 114 in 2011. In 2003, Cancer Control Act was introduced with all reporting hospitals mandated to submit cancer patient information to the cancer registry. To ensure quality of cancer registries and enhancing the quality of cancer registry data, Taiwan Society of Cancer Registry was established in 2006, conducting random medical record review to ensure data accuracy since 2010. TCR data from 2000 through 2018 will be used for this study. | | |
| Study size: | Based on the result of study by Wedzicha JA, et al, (where at least 25% of the patients in the Tio/Olo group have a first moderate or severe exacerbation at 127 days [95% CI, 107 to 149] and in ICS/LABA group at 87 days [95% CI, 81 to 103] (HR = 0.78, [95% CI 0.70 to 0.86])), we assume that at least 25% of patients in the ICS/LABA experienced a first moderate or severe COPD exacerbation at 103 days and the HR of Tio/Olo to LABA/ICS is 0.9. For a study duration of 6 years, a total of 4978 patients (2489 patients each arm) are needed to detect the difference between the two arms with 2-sided alpha of 0.05 and 90% power | | |
| Data analysis: | All variables, including patient characteristics, baseline measures, and outcomes, will be analysed descriptively. All analyses will be presented for each exposure group (Tio+Olo vs LABA/ICS) overall. We will first describe formation of the study cohort. Patient characteristics at baseline in patients treated with Tio+Olo and patients treated with LABA/ICS will be described separately using standard descriptive statistics after propensity score matching. Absolute standardized differences (ASDs) will be used to compare the characteristics between the two groups after propensity score matching, in which a >0.1 ASD indicates a meaningful difference. | | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of same and | | | |
|---|---|---|---|
| Name of company: Boehringer Ingelheim | 1 | | |
| Name of finished me | | | |
| product: | dicinal | | |
| Spiolto Respimat | | | |
| Name of active ingre | | | |
| Tiotropium + Olodate | erol | | |
| {R03AL06} | | | |
| Protocol date: | Study | Version/Revision: | Version/Revision date: |
| 110totol unter | number: | V OI SIOII/ILO VISIOII | v er stom tte vision dave. |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| | annualized rate of exposed group re | ate of moderate or severe COPE<br>of prescriptions of rescue medical<br>elative to LABA/ICS group, alo<br>derived using negative binomia | ations, ratio of Tio+Olo –<br>ng with 95% confidence |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal product: Spiolto Respimat | | | |
| Name of active ingre<br>Tiotropium + Olodate<br>{R03AL06} | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 23 May 2022 | 1237-0110 | 1.0 | NA |
| Milestones: | IRB/IEC approval: 22-Oct-2020 Feasibility assessment: 2020. Q3 EU PAS Registration: 01-Jun-2022 Full analysis: Data Access: 15-Jun-2022 Complete data analysis: 30-Aug-2022 Final report of study results: 15-Oct-2022 Publications timeline: Abstract: 2023 ATS. | | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

# 5. AMENDMENTS AND UPDATES

None

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

## 6. MILESTONES

| Milestone | Planned Date |
|-------------------------------|----------------------|
| IRB/IEC approval | Oct 2020 (completed) |
| Feasibility assessment | Oct 2020 (completed) |
| EU PAS Registration | 01/Jun/2022 |
| Full analysis | |
| Data Access | 15/Jun/2022 |
| Complete data analysis | 30/Aug/2022 |
| Final report of study results | 15/Oct/2022 |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

## 7. RATIONALE AND BACKGROUND

COPD is a leading cause of morbidity and mortality throughout the world. Long-acting bronchodilator medications, which include long-acting β2-agonists (LABAs) and the long-acting muscarinic antagonists (LAMAs) such as tiotropium, are the central maintenance therapy to the management of COPD, with inhaled corticosteroids (ICSs) added with increasing severity. The up-to-date GOLD guideline recommends to initiate ICS/LABA in patients with high blood eosinophils level and frequent exacerbation history[P21-01394]. However, ICS containing therapy has been widely used inappropriately in real world practice.

The role of ICS in COPD has been debated for decades and studies have been conducted to investigate the effect of ICS-containing therapy in patients with COPD. INSPIRE [P07-11820] study indicated that ICS/LABA and tiotropium showed similar effects on the reduction of exacerbations, while the risk of pneumonia was higher in the ICS/LABA group. And the FLAME [P16-05628] study showed LAMA/LABA was superior to ICS/LABA in terms of exacerbation prevention, while in some newly published data focusing on FDC triple therapy showing reversed results.

With more and more fixed dose combination medications, i.e. LAMA/LABA, ICS/LABA/LAMA, approved and prescribed in recent years, it is of clinical interests to understand the effectiveness and safety profile of these therapies in real world settings.

The aim of this real world study is to assess effectiveness and safety profile between tiotropium/olodaterol (Tio/Olo) and ICS/LABA. The primary outcome of the study will be time to first moderate or severe COPD exacerbations. Other outcomes include time to ICS/LABA/LAMA escalation, rate of escalation to triple therapy, pneumonia and rescue medication use.

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

# 8. RESEARCH QUESTION AND OBJECTIVES

# Primary objective:

• To compare time to the first moderate or severe COPD exacerbations between initiators of Tio/Olo and ICS/LABA in a real world setting;

## Secondary objectives:

- To compare time to escalation to triple therapy between initiators of Tio/Olo and ICS/LABA;
- To compare the rate of escalation to triple therapy between initiators of Tio/Olo and ICS/LABA;
- To compare the time to first hospitalization for community-acquired pneumonia between initiators of Tio/Olo and ICS/LABA;
- To compare the number of prescriptions of rescue medication between initiators of Tio/Olo and ICS/LABA;
- To compare the annualized rate of moderate or severe COPD exacerbation between initiators of Tio/Olo and ICS/LABA..

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

#### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This study will be a non-interventional cohort study based on existing data (NISed).

The aim of this real world study is to assess effectiveness and safety profile between tiotropium/olodaterol (Tio/Olo) and ICS/LABA. The primary outcome of the study will be time to the first moderate or severe COPD exacerbations. Other outcomes include time to ICS/LABA/LAMA escalation, rate of escalation to triple therapy, pneumonia and rescue medication use.

#### 9.2 SETTING

## 9.2.1 Study sites

Data used in this study will come from the Taiwan National Health Insurance (NHI) claims data between 2014 and 2019.

## 9.2.2 Study population

#### Inclusion criteria:

- At least oneprescriptions for Tio/Olo combined inhaler or a LABA/ICS combined inhaler between 1<sup>st</sup> January 2014 and 31<sup>st</sup> December 2019.
  - a) The first dispensing of either Tio/Olo or LABA/ICS combined inhaler will be defined as the index date;
  - b) For the main analyses, only fixed dose combination (FDC) inhalers will be included.
- 2. Aged  $\geq$  40 years on the index date
- 3. At least one diagnosis of COPD at any time prior to or on the index date;
- At least one year of continuous medical and health insurance plan prior to the index date will be required to allow for a look-back period for the covariates and identification of new use of the study drugs;
- 5. At least one record in the health insurance system database;

#### Exclusion criteria:

- 1. Any use of Tio/Olo, ICS/LABA, or ICS/LAMA/LABA in free or fixed form for one year prior to the index date;
- Individuals with asthma, allergic rhinitis, lung cancer, interstitial lung disease, or lung transplant identified at any time prior to the index date

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

For the analysis of the primary outcome, individuals will be followed up from the index date until the earliest of the date of: the follows, whichever first 1) moderate or severe COPD exacerbation; 2) disenrollment; 3) the end of the study period; 4) death; 5) discontinuation of the index drug use as a lapse of 1.5 months without subsequent prescription (except for switching from the index ICS/LABA to a different ICS/LABA); 6) adding ICS mono on top of Tio/Olo, or adding LAMA momo on top of the index ICS/LABA

#### 9.2.3 Study visits

Not applicable

#### 9.2.4 Study discontinuation

Boehringer Ingelheim reserves the right to discontinue the study at any time for the following reasons:

1. Violation of Good Pharmacoepidemiology Practice (GPP), the study protocol, or the contract by a study site, investigator or research collaborator, disturbing the appropriate conduct of the study

#### 9.3 VARIABLES

#### 9.3.1 Exposures

Exposure of this study is defined as new initiation of Tiotropium/Olodaterol, or ICS/LABA during the study period.

#### 9.3.2 Outcomes

#### 9.3.2.1 Primary outcomes

- Outcome type: Primary
- Outcome Name: Time to the first moderate or severe COPD exacerbations after index date
- Time Frame: 2014~2019Safety Issue (Yes/No): No

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

#### 9.3.2.2 Secondary outcomes

- Outcome type: Secondary

- Outcome Name: Time to triple therapy escalation after index date

Time Frame: 2014~2019Safety Issue (Yes/No): No

- Outcome type: Secondary

- Outcome Name: Incidence rate of triple therapy initiation (first event per patient)

Time Frame: 2014~2019Safety Issue (Yes/No): No

- Outcome type: Secondary

- Outcome Name: Time to the first hospitalization for community-acquired pneumonia after entry

Time Frame: 2014~2019Safety Issue (Yes/No): No

- Outcome type: Secondary

- Outcome Name: Annualized rate of prescriptions of rescue medications after the index date

- Calculation: annualized rate=number of prescriptions/total patient year at risk=number of prescriptions per patient year

Time Frame: 2014~2019Safety Issue (Yes/No): No

- Outcome type: Secondary

- Outcome Name: Annualized rate of moderate or severe COPD exacerbation after the index date

- Calculation: annualized rate=number of moderate or severe COPD exacerbations/total patient year at risk=number of exacerbations per patient year

Time Frame: 2014~2019Safety Issue (Yes/No): No

#### 9.3.3 Covariates

Demographic characteristics and cohort entry information:

Sex

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

- Age
- Calendar year of cohort entry
- Season of index date (winter, spring, summer, fall)

Additional, the following clinical characteristics will be measured during the 1 year pre-index baseline period:

#### Previous COPD treatments

- ➤ LAMA monotherapy
- ➤ LABA monotherapy
- > ICS monotherapy
- ➤ LAMA/ICS combination therapy

Use of other respiratory drugs

- Mucolytics
- > Theophylline
- ➤ Short-acting beta-agonists
- > Short-acting muscarinic antagonists
- Previous acute COPD exacerbation (measured both 12 months and in the 30 days prior to cohort entry), categorized as 0, 1 or 2+.
  - ➤ All exacerbations (Moderate+Severe)
  - An outpatient visit with a diagnosis code for COPD in any field + a prescription for an oral corticosteroid or an antibiotic for respiratory infections (Moderate)
  - ➤ Hospitalizations or emergency room visits with a primary diagnosis for COPD (Severe)
- Hospitalizations caused by exacerbation of COPD in 12 months prior to the index date:
  - **>** 0;
  - **>** 1;
  - **>** 2+;
- all-cause hospitalizations in 12 months prior to index date:
  - > 0;
  - **>** 1;
  - **>** 2+;
- Comorbidities:
  - > Cardiovascular disease
  - > Cerebrovascular disease
  - Diabetes
  - > Chronic kidney disease
  - > Pneumonia
  - > Cancer
  - Cirrhosis

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

- Charlson Comorbidity Index (CCI)
- History of medications dispensed in the 12 months before or on the index date will be identified from the pharmacy dispensing history:
  - > Cardiovascular drugs:

Antihypertensives

Antiarrhythmics

**Nitrates** 

heart failure medications

- ➤ Lipid-lowering medications
- ➤ Blood glucose-lowering medications
- ➤ Anticoagulants and antiplatelet agents
- > Antibiotics
- ➤ Antineoplastic agents

#### COPD severity

The definition of the severity of COPD in this study was developed based on the information in previous studies, GOLD recommendations and clinical practice in Taiwan, see below. Patients who fulfil criteria for more than one category will be classified as being in the most severe category.

## Criteria of COPD severity:

➤ Mild:

Naïve to COPD treatment, or at least one dispensing of the following categories of medications either alone or in combination: 1) SABA or SAMA or SABA+SAMA, 2) LAMA or LABA monotherapy, 3) theophylline or mucolytics, in the 12 months before the index date;

#### ➤ Moderate:

At least one dispensing of LAMA + LABA in the 12 months before the index date;

#### > Severe:

Occurrence of at least one of the following events in the 12 months before the index date:

- Hospitalisation for COPD
- Recorded diagnosis of pneumonia
- Second course of antibiotics for respiratory tract infections
- Second course of systemic corticosteroids for the treatment of COPD exacerbation
- Two diagnoses of COPD exacerbation without hospitalisation

#### ➤ Very severe:

Occurrence of at least one of the following events in the 12 months before the index date unless other time period is specified:

- Dispensed oxygen therapy
- Dispensed nebuliser therapy

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

#### 9.4 DATA SOURCES

Data used in this study will come from the Taiwan National Health Insurance (NHI) claims data between 2014 and 2019.

Data sources include Taiwan NHI, Taiwan cancer registry (TCR) and Taiwan Mortality Data. Taiwan Department of Statistics, Ministry of Health and Welfare is the unit designated by the government to manage health and social welfare statistical databases, and to develop data platform for academic research. Through the services provided by the Health and Welfare Data Science Center (HWDSC) of the Department of Statistics, researchers may access a wide range of health and welfare data, including claims, mortality (with cause of death) and Taiwan Cancer Registry (TCR). The HWDSC staff encrypt the national ID for all individuals according to a secure encryption algorithm that is not made known to the public. The encrypted ID is unique for all individuals and will be used for linkage between databases.

#### (a) National Health Insurance claims data

Taiwan National Health Insurance (NHI) started in 1995 and is a publicly funded single payer health insurance program for all residents. Health insurance for individuals is required by law and coverage is more than 99%. The majority healthcare providers in Taiwan contract with the National Health Insurance Agency in Taiwan to provide a wide range of medical services. Geographic locations of health care claims are broadly classified into 6 regions in Taiwan. Salary range, which serves as the basis for enrollees' premium calculation, can serve as a proxy indicator for socioeconomic status. Bundled payment according to the Diagnosis-Related Group system only applies in limited number of disease conditions, therefore detailed drug use information during hospitalization is also available. An added advantage of the NHI data source is the low membership turnover rate, which is particularly important for longterm follow-up study. NHI claims were based on International Classification of Disease, ninth revision, clinical modification (ICD-9-CM) codes till the end of 2015, and then switched to International Classification of Disease, tenth revision, clinical modification (ICD-10-CM) codes after 2016. Specific NHI data column please see file "column note in TW NHI 20210824" [No document #] in the database (confidential and only can be accessed by PI).

#### (b) Mortality data

The household registration system in Taiwan maintain birth, marital status, and death information and is administrated by the Department of Household Registration, Ministry of the Interior. Death certificates are collected through this system and transferred to the Ministry of Housing and Works (MOHW) for coding of cause of death and maintenance of the mortality database. The cause of death was coded in the ICD-9-CM format from 1990 to 2009, and in ICD-10-CM format from 2010 to 2019. This study will use the cause of death files in years 2012-2019, primarily focusing on the date of death of study subjects.

#### (c) Taiwan Cancer Registry data

In Taiwan, the population-based cancer registry was founded in 1979. Since then, the registry collected basic information, referred to the "20 items short-form system," on incident cancer cases (including cancer-in-situ) within one year after the initial diagnosis from hospitals with more than 50-bed capacity throughout the country. Recorded items include date of birth, gender, time and method of diagnosis, cancer site and morphology, treatment summary and

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

death. From 2002 onward, a "long-form" system was established to collect more detailed information of cancer staging, treatment and follow-up data from hospitals with more than 500 new cancer cases diagnosed annually. The number of recorded items increased from 20 to 65 in 2002, further to 95 in 2007, and to 114 in 2011. In 2003, Cancer Control Act was introduced with all reporting hospitals mandated to submit cancer patient information to the cancer registry. To ensure quality of cancer registries and enhancing the quality of cancer registry data, Taiwan Society of Cancer Registry was established in 2006, conducting random medical record review to ensure data accuracy since 2010. TCR data from 2000 through 2018 will be used for this study.

#### 9.5 STUDY SIZE

Based on the result of study by Wedzicha JA, et al, [P16-05628] (where at least 25% of the patients in the Tio/Olo group have a first moderate or severe exacerbation at 127 days [95% CI, 107 to 149] and in ICS/LABA group at 87 days [95% CI, 81 to 103] (HR = 0.78, [95% CI 0.70 to 0.86])), we assume that at least 25% of patients in the ICS/LABA experienced a first moderate or severe COPD exacerbation at 103 days and the HR of Tio/Olo to LABA/ICS is 0.9. For a study duration of 6 years, a total of 4978 patients (2489 patients each arm) are needed to detect the difference between the two arms with 2-sided alpha of 0.05 and 90% power

## 9.6 DATA MANAGEMENT

Full details of the data management plan are documented in a separate NIS-Data Management and Review Plan (NIS-DMRP).

## 9.7 DATA ANALYSIS

Full details of the statistical analysis will be documented in the SEAP, which will be finalized before the end of data collection.

## 9.7.1 Main analysis

All variables, including patient characteristics, baseline measures, and outcomes, will be analyzed descriptively.

- For all analyses, variables will be reported as follows: Continuous variables (e.g., age) will be presented as means (with standard deviation, SD) and/or medians (with interquartile range, IQR), minimum, maximum.
- Categorical variables (e.g., sex) will be presented as absolute and relative frequencies.

All analyses will be presented for each treatment group (Tio+Olo vs LABA/ICS) overall. We will first describe formation of the study cohort. Propensity score matching will be used to balance the baseline characteristics of patients in the two treatment groups. The covariates used to calculate the propensity score would be specified in the SEAP. All the analyses will be performed on patients after propensity score matching. Patient characteristics at baseline in patients treated with Tio+Olo and patients treated with LABA/ICS will be described separately using standard descriptive statistics after propensity score matching. Absolute standardized differences (ASDs) will be used to compare the characteristics between the two

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

groups after propensity score matching, in which a >0.1 ASD indicates a meaningful difference.

For the analysis of the primary outcome, individuals will be followed up from the index date until the first moderate or severe COPD exacerbation. The data after the earliest date of the following would be censored: 1) disenrollment; 2) the end of the study period; 3) death; 4) discontinuation of the index drug (except for switching from the index ICS/LABA to a different ICS/LABA); 5) escalation to triple therapies (ICS/LAMA/LABA free or fix dose combination). Cox proportional hazard regression model will be used to compare the time to event between the two treatment groups, while accounting for the potential baseline differences between them. Other known predictors will also be included in the model as covariates. It will provide an estimate of the hazard ratio (HR) of time to the first moderate or severe COPD exacerbation associated with Tio+Olo use relative to LABA/ICS use, along with 95% confidence intervals (CI). The analysis will be on-treatment.

The analysis of the secondary objectives related to time to triple therapy escalation, time to first hospitalization for community-acquired pneumonia, will use a Cox proportional hazard regression model with an as-treated approach, similar to that of the primary analysis. The estimate of hazard ratio (HR) of time to triple therapy escalation and first hospitalization for community-acquired pneumonia associated with Tio+Olo use relative to LABA/ICS use, along with 95% confidence intervals (CI) will be provided. For the analysis of these time-to-event outcomes, patients will be followed up until until the earliest of the date of the follows, whichever happened first 1) outcome event of interest; 2) disenrollment; 3) the end of the study period; 4) death; 5) discontinuation of the index drug (except for switching from the index ICS/LABA to a different ICS/LABA).

For incidence rate of triple therapy initiation (first event per patient), annualized rate of moderate or severe COPD exacerbations, and annualized number of prescriptions of rescue medications will be calculated by cohort.

For continuous and categorical variables, we will use standard descriptive statistics to describe. For incidence rates, it will be calculated for each cohort as follows: Incidence rate among the Tio+Olo cohort = (total number of patients in the Tio+Olo cohort experiencing an event of interest for the first time during the given time period) / (total person-time at risk from current use of Tio+Olo during the given period)

Incidence rate among the comparison cohort = (total number of patients in the comparator LABA/ICS cohort experiencing an event of interest for the first time during the given time period) / (total person-time at risk from current use of comparator LABA/ICS during the given period)

The incidence rate ratio (IRR) and incidence difference for the outcome in the Tio+Olo - exposed group relative to that in the comparator group will be derived as follows:

Incidence rate ratio = incidence rate from the Tio+Olo cohort divided by the incidence rate from the matched comparator cohort.

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

Incidence difference = incidence rate from the Tio+Olo cohort – incidence rate from the matched comparator cohort

The IRRs will be calculated. Incidence differences and their 95% confidence intervals will also be derived.

For annualized rates, it will be calculated for each cohort as follows:

Annualized rate among the Tio+Olo cohort = (total number of events in the Tio+Olo cohort during the given time period) / (total person-time at risk from current use of Tio+Olo during the given period)

Annualized rate among the comparison cohort = (total number of events in the comparator LABA/ICS cohort during the given time period) / (total person-time at risk from current use of comparator LABA/ICS during the given period)

The incidence rate ratio (IRR) for the triple therapy initiation in the Tio+Olo - exposed group relative to that in the comparator group, along with 95% confidence intervals will be derived using negative binomial model.

For annualized rate of moderate or severe COPD exacerbations and annualized number of prescriptions of rescue medications, the ratio of Tio+Olo – exposed group relative to LABA/ICS group, along with 95% confidence intervals will be derived using negative binomial model.



#### 9.7.3 Safety Analysis

Based on current guidelines from the International Society for Pharmacoepidemiology [R11-4318] and the EMA [R13-1970], non-interventional studies such as the one described in this propotol, conducted using health care records, do not require expedited reporting of suspected adverse events/reactions. Specifically, as stated in section VI.C.1.2.1 of Guideline on Good Pharmacovigilance Practices (GVP), Module VI – Management and Reporting of Adverse Reactions to Medicinal Products, for non-interventional study designs, which are based on use of secondary data, reporting of adverse reactions is not required.

#### 9.8 QUALITY CONTROL

The study will strictly follow relevant BI SOPs. In addition, this study will follow key elements of the Guideline for Good Pharmacoepidemiology Practices (GPP). The statistical

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

analytic approach will be reviewed/repeated by a second analyst to ensure quality control. The study report will be reviewed, approved and archived per BI SOP

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

Some important potential confounders are not available in the Taiwan NHI dataset. For example, pulmonary function data and duration of COPD may not be available in the data set. These variables will not be calculated so there might be confounding bias in the study. The definition for COPD severity was developed based on the previous evidence, treatment guideline and the clinical practice in Taiwan to reduce the bias.

COPD patients concomitant with asthma may be different from COPD patients without asthma in terms of the disease natural course, treatment regimen, and response to drugs. Therefore, COPD patients concomitant with asthma will be excluded from the primary analysis. Previous studies suggested that there might be misdiagnosis between COPD and asthma. To further exclude potential asthma patients,

In a database study like this, we can only rely on the available information to define outcomes, exposure and covariates. There will be misclassification of study variables. In the analyses, whenever possible, validated algorithm will be used to reduce misclassifications.

#### 9.10 OTHER ASPECTS

#### 9.10.1 Data quality assurance

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by Institutional Review Board (IRBs) / Independent Ethics Committee (IECs) or by regulatory authorities. The quality assurance auditor will have access to the investigator's study-related files and correspondence.

#### 9.10.2 Study records

#### 9.10.2.1 Source documents

#### Not applicable

Data are provided by Health and Welfare Data Science Center, Ministry of Health and Welfare, Taiwan. Data access was only available through dedicated data analysis areas within the Ministry. Individual level data are not allowed to be brought outside of the Ministry.

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

9.10.2.2 Direct access to source data and documents

Not applicable.

Data are provided by Health and Welfare Data Science Center, Ministry of Health and Welfare, Taiwan. Data access was only available through dedicated data analysis areas within the Ministry. Individual level data are not allowed to be brought outside of the Ministry.

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

## 10. PROTECTION OF HUMAN SUBJECTS

The study will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, Guidelines for Good Pharmacoepidemiology Practice (GPP), and the relevant BI Standard Operating Procedures (SOPs).

# 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This NIS will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB)/Independent Ethics Committee (IEC) and Competent Authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments

#### 10.2 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Data generated as a result of the study need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB/IEC and the regulatory authorities.

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

#### 11.1 DEFINITIONS OF ADVERSE EVENTS

Not applicable

# 11.2 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING

Not applicable based on secondary use of data without any potential that any employee of BI or agent working on behalf of BI will access individually identifiable patient data.

This study is a non-interventional study based on secondary data without involving review or analysis of any individual patient level data. The data is extracted and analyzed in an aggregate manner.

## 11.3 REPORTING TO HEALTH AUTHORITIES

This study is a non-interventional study based on secondary data, which will not involve individual medical record review. Therefore, no AE collection of this study will be performed and reported to Chinese regulatory authorities.

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.
NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

#### 13. REFERENCES

#### 13.1 PUBLISHED REFERENCES

**P21-01394** Global initiative for chronic obstructive lung disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease (2021 REPORT). https://goldcopd.org/goldreports/.

**P07-11820** Wedzicha JA et al. The prevention of COPD exacerbations by salmeterol/fluticasone propionate or tiotropium bromide. Am J Respir Crit Care Med.2008;177:19-26.

**P16-05628** Wedzicha J A, et al. Indacaterol–Glycopyrronium versus Salmeterol–Fluticasone for COPD. N Engl J Med, 2016, 2016(374): 2222-2234

**R11-4318** Guidelines for Good Pharmacoepidemiology Practices (GPP) (revision 3: June 2015). Guidelines for Good Pharmacoepidemiology Practices (GPP) - International Society for Pharmacoepidemiology (access date: 1st March 2022); International Society for Pharmacoepidemiology (ISPE); 2015.

R13-1970 European Medicines Agency (EMA), Heads of Medicines Agencies (HMA); Guideline on good pharmacovigilance practices (GVP): module VI - management and reporting of adverse reactions to medicinal products (28 July 2017 EMA/873138/2011 Rev 2). Guideline on good pharmacovigilance practices (GVP) - Module VI – Collection, management and submission of reports of suspected adverse reactions to medicinal products (Rev 2) (europa.eu) (access date: 1st March 2022); European Medicines Agency (EMA), Heads of Medicines Agencies (HMA); 2017.

#### 13.2 UNPUBLISHED REFERENCES

**No document** # Taiwan National Health Insurance, *column\_note\_in\_TW\_NHI\_20210824*. 24 Aug 2021

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

#### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

| Number | Document<br>Reference Number | Date | Title |
|--------|------------------------------|------|-------|
| None | | | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

#### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

#### Study title:

**EU PAS Register® number:** 

Effectiveness of Maintenance Treatment with Tiotropium + Olodaterol in Comparison to Inhaled Corticosteroids + Long-acting  $\beta 2$  agonists in COPD patients in Taiwan: a non-interventional study based on the Taiwan National Health Insurance (NHI) data.

| Section 1: Milestones | Yes | No | N/A | Section Numbe |
|---|---|---|---|---|
| 1.1 Does the protocol specify timelines for | | | | |
| 1.1.1 Start of data collection <sup>1</sup> | | | $\boxtimes$ | |
| 1.1.2 End of data collection <sup>2</sup> | | | $\boxtimes$ | |
| 1.1.3 Progress report(s) | | | $\boxtimes$ | |
| 1.1.4 Interim report(s) | | | $\boxtimes$ | |
| 1.1.5 Registration in the EU PAS<br>Register® | | | | |
| 1.1.6 Final report of study results. | $\boxtimes$ | | | <u>6</u> |

| Section 2: Research question | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|
| 2.1 Does the formulation of the research question and objectives clearly explain: | | | | |
| 2.1.1 Why the study is conducted? (e.g. to address an important public health concern, a risk identified in the risk management plan, an emerging safety issue) | | | | 7 |
| 2.1.2 The objective(s) of the study? | $\boxtimes$ | | | <u>8</u> |
| 2.1.3 The target population? (i.e. population or<br>subgroup to whom the study results are intended to<br>be generalised) | | | | 9.2.2 |
| 2.1.4 Which hypothesis(-es) is (are) to be tested? | | | | |
| 2.1.5 If applicable, that there is no a priori hypothesis? | | | | |

\_

<sup>1</sup> Date from which information on the first study is first recorded in the study dataset or, in the case of secondary use of data, the date from which data extraction starts.

<sup>2</sup> Date from which the analytical dataset is completely available.

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| nmen | ts: | | | | |
|---|---|---|---|---|---|
| Sect | ion 3: Study design | Yes | No | N/A | Sectio<br>Numb |
| 3.1 | Is the study design described? (e.g. cohort, case-control, cross-sectional, other design) | $\boxtimes$ | | | 9. |
| 3.2 | Does the protocol specify whether the study is based on primary, secondary or combined data collection? | $\boxtimes$ | | | 9.4 |
| 3.3 | Does the protocol specify measures of occurrence? (e.g., rate, risk, prevalence) | $\boxtimes$ | | | 9.3 |
| 3.4 | Does the protocol specify measure(s) of association? (e.g. risk, odds ratio, excess risk, rate ratio, hazard ratio, risk/rate difference, number needed to harm (NNH)) | $\boxtimes$ | | | 9.7 |
| 3.5 | Does the protocol describe the approach for the collection and reporting of adverse events/adverse reactions? (e.g. adverse events that will not be collected in case of primary data collection) | | | | 11 |
| nmen | ts: | | | | |
| | ion 4: Source and study<br><u>Jlations</u> | Ye<br>s | No | N/A | Sectio<br>Numb |
| 4.1 | Is the source population described? | | | | 9.4 |
| 4.2 | Is the planned study population defined in terms of: | | | | |
| 4.2.1 | Study time period | | | | 9.2 |
| 4.2.2 | 2 Age and sex | | | | 9.2 |
| 4.2.3 | 3 Country of origin | | | | 9.4 |
| 4.2.4 | Disease/indication | | | | 9.2 |
| 4.2.5 | Duration of follow-up | | | | 9.2 |
| 4.2 | Does the protocol define how the | | | | 9.2 |
| 4.3 | study population will be sampled from<br>the source population? (e.g. event or<br>inclusion/exclusion criteria) | | | | 3.2 |
| 4.3<br>nmen | the source population? (e.g. event or inclusion/exclusion criteria) | | | | 5.2 |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| | tion 5: Exposure definition and surement | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 5.1 | Does the protocol describe how the study exposure is defined and measured? (e.g. operational details for defining and categorising exposure, measurement of dose and duration of drug exposure) | | | | 9.3.1 |
| 5.2 | Does the protocol address the validity of the exposure measurement? (e.g. precision, accuracy, use of validation substudy) | | | | |
| 5.3 | Is exposure categorised according to time windows? | | | $\boxtimes$ | |
| 5.4<br>(e.g. | Is intensity of exposure addressed? dose, duration) | | $\boxtimes$ | | |
| 5.5 | Is exposure categorised based on biological mechanism of action and taking into account the pharmacokinetics and pharmacodynamics of the drug? | | | $\boxtimes$ | |
| 5.6<br>mmen | Is (are) (an) appropriate comparator(s) identified? | | | | 9.1 |
| mmen<br>Sect | comparator(s) identified? hts: tion 6: Outcome definition and | Yes | No | N/A | Section |
| mmen<br>Sect | comparator(s) identified? | | No | N/A | Section<br>Number |
| mmen<br>Sect<br>mea | comparator(s) identified? Ints: Ition 6: Outcome definition and insurement Does the protocol specify the primary and secondary (if applicable) outcome(s) | Yes | No | N/A | Section<br>Number |
| Sect<br>mea<br>6.1 | comparator(s) identified? Ints: Ition 6: Outcome definition and insurement Does the protocol specify the primary and secondary (if applicable) outcome(s) to be investigated? Does the protocol describe how the | Yes | No | N/A | 9.1<br>Section<br>Number<br>9.3.2 |
| Sect mea 6.1 | comparator(s) identified? Ints: Ition 6: Outcome definition and issurement Does the protocol specify the primary and secondary (if applicable) outcome(s) to be investigated? Does the protocol describe how the outcomes are defined and measured? Does the protocol address the validity of outcome measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, use of validation sub- | Yes | | N/A | Section<br>Number |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Secti | on 7: Bias | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|---|
| 7.1 | Does the protocol address ways to measure confounding? (e.g. confounding by indication) | $\boxtimes$ | | | 9.7.1 |
| 7.2 | Does the protocol address selection bias? (e.g. healthy user/adherer bias) | | $\boxtimes$ | | |
| | Does the protocol address information bias? (e.g. misclassification of exposure and outcomes, time-related bias) | | | | 9.9 |
| Comment | CS: | | | | |
| Section | 8: Effect measure modification | Yes | No | N/A | Section<br>Number |
| 8.1 | Does the protocol address effect<br>modifiers? (e.g. collection of data on known<br>effect modifiers, sub-group analyses,<br>anticipated direction of effect) | | | | |
| Comment | CS: | | | | |
| <u>Secti</u> | on 9: Data sources | Yes | No | N/A | Section<br>Number |
| | Does the protocol describe the data source(s) used in the study for the ascertainment of: | | | | |
| ger | Exposure? (e.g. pharmacy dispensing, neral practice prescribing, claims data, selfort, face-to-face interview) | | | | <u>9.4</u> |
| ma<br>inte | Outcomes? (e.g. clinical records, laboratory rkers or values, claims data, self-report, patient erview including scales and questionnaires, vital tistics) | | | | <u>9.4</u> |
| 9.1.3 | Covariates and other characteristics? | | | | <u>9.4</u> |
| | Does the protocol describe the information available from the data source(s) on: | | | | |
| qua | Exposure? (e.g. date of dispensing, drug antity, dose, number of days of supply scription, daily dosage, prescriber) | | | | <u>9.4</u> |
| | Outcomes? (e.g. date of occurrence, multiple ent, severity measures related to event) | | | | 9.4 |
| (e. | Covariates and other characteristics? g. age, sex, clinical and drug use history, corbidity, co-medications, lifestyle) | $\boxtimes$ | | | <u>9.4</u> |
| 9.3 | Is a coding system described for: | | | | |
| Ana | Exposure? (e.g. WHO Drug Dictionary, atomical Therapeutic Chemical (ATC) ssification System) | | | | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Proprietary confidential | information © 2022 Boehringer Ingelheim Inte | ernational Gmbl | H or one of | or more of its | affiliated |
|---|---|---|---|---|---|
| Section 9: Data | <u>sources</u> | Yes | No | N/A | Section<br>Number |
| | (e.g. International Classification<br>Medical Dictionary for Regulatory<br>A)) | | | | 9.4 |
| 9.3.3 Covariates | and other characteristics? | | | | |
| | method between data cribed? (e.g. based on a unique her) | | | | 9.4 |
| Comments: | | | | | |
| Specifics will be o | lescribed in SEAP. | | | | |
| Section 10: Ana | lysis plan | Yes | No | N/A | Section<br>Number |
| | istical methods and the heir choice described? | $\boxtimes$ | | | 9.7 |
| 10.2 Is study siz precision es | e and/or statistical<br>stimated? | | | | <u>9.5</u> |
| 10.3 Are descript | tive analyses included? | $\boxtimes$ | | | 9.7.1 |
| 10.4 Are stratifie | d analyses included? | | | | 9.7.2 |
| • | an describe methods for atrol of confounding? | $\boxtimes$ | | | 9.7.1 |
| | an describe methods for atrol of outcome atron? | | $\boxtimes$ | | |
| 10.7 Does the pl<br>handling mi | an describe methods for ssing data? | | $\boxtimes$ | | |
| Comments: | | | | | |
| Section 11: Dat quality control | a management and | Yes | No | N/A | Section<br>Number |
| on data sto | otocol provide information<br>rage? (e.g. software and IT<br>database maintenance and anti-<br>on, archiving) | | | | |
| 11.2 Are method described? | s of quality assurance | | | | <u>9.8</u> |
| | ystem in place for<br>t review of study results? | | | | |
| Comments: | | | | | |

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

| Section 12: Limitations | Yes | No | N/A | Section<br>Number |
|---|---|---|---|---|
| 12.1 Does the protocol discuss the impact on the study results of: | | | | |
| 12.1.1 Selection bias? | $\boxtimes$ | | | <u>9.9</u> |
| 12.1.2 Information bias? | $\boxtimes$ | | | <u>9.9</u> |
| 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). | | | | 9.9 |
| 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | | | | <u>9.5</u> |
| Comments: | | | | |
| Section 13: Ethical/data protection issues | Yes | No | N/A | Section<br>Number |
| 13.1 Have requirements of Ethics Committee/ Institutional Review Board been described? | | | | 9.10.1 |
| 13.2 Has any outcome of an ethical review procedure been addressed? | | | | |
| 13.3 Have data protection requirements been described? | | | | |
| Comments: | | | | |
| Section 14: Amendments and deviations | Yes | No | N/A | Section<br>Number |
| 14.1 Does the protocol include a section to document amendments and deviations? | $\boxtimes$ | | | <u>5</u> |
| Comments: | | | | |
| Section 15: Plans for communication of study results | Yes | No | N/A | Section<br>Number |
| 15.1 Are plans described for communicating study results (e.g. to regulatory authorities)? | $\boxtimes$ | | | <u>12</u> |
| 15.2 Are plans described for disseminating study results externally, including publication? | $\boxtimes$ | | | 12 |

**NIS Protocol** 

BI Study Number: 1237-0110

 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

| IS Protocol | Page 45 of 4 |
|---|---|
| I Study Number: 1237-0110 | c38660249-0 |
| Proprietary confidential information © 2022 Boehringer Ingelhein | International GmbH or one or more of its affiliated |
| Comments: | |
| Name of the main author of the protocol: | |
| | , |
| Date: May 23, 2022 | |
| Name of the main author of the protocol: | |
| Date: May 23, 2022 | |

001-MCS-90-118\_RD-23 (2.0) / Saved on: 02 Jul 2020

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

#### **ANNEX 3. ADDITIONAL INFORMATION**

None

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

#### ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES

The NIS Protocol must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI product(s) | NIS not invo | lving BI product(s) |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi | X | X | X |
| Global TMM / TMMA / TM Market<br>Access | X | X | |
| Global Project Statistician | X | X | |
| Global TM RA | X | | |
| Global PVWG Chair | X | | |
| GPV SC | X | X | X |
| Global CTIS representative | X | | |
| Local Medical Director | X (if local study) | | X |
| Local Head MAcc / HEOR Director | X (if local study) | | X |
| Global TA Head Epi* | X | X | |
| Global TA Head Clinical<br>Development / Medical Affairs /<br>Market Access* | X | X | |
| Global TA Head PV RM* | X | | |
| RWE CoE | X | X | |
| PSTAT / PSTAT-MA<br>(for NISnd only) | X | X | X |
| NIS DM | X | X | X |
| Local Head MA/Clinical<br>Development | | | X (does not apply to<br>NISed without chart<br>abstraction) |

<sup>\*</sup> After review by Global TM for function

NIS Protocol  BI Study Number: 1237-0110 c38660249-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated

Study Title: Effectiveness of Maintenance Treatment with Tiotropium + Olodaterol in Comparison to Inhaled Corticosteroids + Long-acting  $\beta 2$  agonists in COPD patients in Taiwan: a non-interventional study based on the Taiwan National Health Insurance (NHI) data.

**Study Number: 1237-0110** 

**Protocol Version:1.0** 

I herewith certify that I agree to the content of the study protocol and to all documents referenced in the study protocol.

Note: Please insert respective signatories with regard to the SOP.

| Position: | Name/Date: | Signature: |
|-----------|------------|------------|
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |